CLINICAL TRIAL: NCT04429295
Title: Immunogenicity and Safety of a DTwP-HepB-Hib-IPV (Shan6™) Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers in Thailand
Brief Title: Study of DTwP-HepB-Hib-IPV (SHAN6™) Vaccine Administered Concomitantly With Routine Pediatric Vaccines to Healthy Infants and Toddlers in Thailand
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SH600009; U1111-1233-9694 (Other: UTN)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pertussis Immunisation; Diphtheria Immunisation; Polio Immunisation; Hepatitis B Immunisation; Haemophilus Influenzae Type B Immunisation; Tetanus Immunisation; Rotavirus Immunisation; Pneumococcal Immunisation
MeSH Terms: interventions — Diphtheria Toxoid; Tetanus Toxoid; Hepatitis B Surface Antigens; Poliovirus Vaccine, Inactivated; RIX4414 vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Intervention regimen (Experimental): SHAN6™ + routine pediatric vaccines pneumococcal 13-valent conjugate vaccine [PCV] [Prevnar 13®] and oral rotavirus vaccine [ORV-1] [Rotarix™] at age of 2, 4 months; SHAN6™ + Prevnar 13® at age of 6 months; SHAN6™ administered alone as a booster dose at age of 15-18 months
  Interventions: Biological: DTwP-HepB-Hib-IPV hexavalent vaccine (Diphtheria toxoid, Tetanus toxoid, whole cell pertussis, Hepatitis B surface antigen (HBsAg), Haemophilus influenzae type b, inactivated poliovirus); Biological: Human Rotavirus, live attenuated; Biological: Pneumococcal polysaccharide conjugate vaccine (13-valent, adsorbed)
- Group B - Control regimen (Active Comparator): SHAN5™ + bivalent oral polio vaccine (bOPV), co-administered with Prevnar 13® and Rotarix™ at 2, 4 months of age and with inactivated polio vaccine [IPV] at 4 months of age; SHAN5™ + bOPV, co-administered with Prevnar 13® at 6 months of age SHAN6™ administered alone as a booster dose at 15-18 months of age
  Interventions: Biological: DTwP-HepB-Hib-IPV hexavalent vaccine (Diphtheria toxoid, Tetanus toxoid, whole cell pertussis, Hepatitis B surface antigen (HBsAg), Haemophilus influenzae type b, inactivated poliovirus); Biological: DTwP-HepB-Hib pentavalent vaccine (Diphtheria toxoid, Tetanus toxoid, whole cell pertussis, Hepatitis B surface antigen (HBsAg), Haemophilus influenzae type b); Biological: Inactivated Poliomyelitis Vaccine; Biological: Poliomyelitis Vaccine bivalent types 1 and 3; Biological: Human Rotavirus, live attenuated; Biological: Pneumococcal polysaccharide conjugate vaccine (13-valent, adsorbed)

INTERVENTIONS:
Biological: DTwP-HepB-Hib-IPV hexavalent vaccine (Diphtheria toxoid, Tetanus toxoid, whole cell pertussis, Hepatitis B surface antigen (HBsAg), Haemophilus influenzae type b, inactivated poliovirus) — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Other Names: SHAN6™
Biological: DTwP-HepB-Hib pentavalent vaccine (Diphtheria toxoid, Tetanus toxoid, whole cell pertussis, Hepatitis B surface antigen (HBsAg), Haemophilus influenzae type b) — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Other Names: SHAN5™
  Arms: Group B - Control regimen
Biological: Inactivated Poliomyelitis Vaccine — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Other Names: IMOVAX Polio
  Arms: Group B - Control regimen
Biological: Poliomyelitis Vaccine bivalent types 1 and 3 — Pharmaceutical form:Oral suspension Route of administration: Oral
  Arms: Group B - Control regimen
Biological: Human Rotavirus, live attenuated — Pharmaceutical form:Oral suspension Route of administration: Oral
  Other Names: Rotarix™
Biological: Pneumococcal polysaccharide conjugate vaccine (13-valent, adsorbed) — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Other Names: Prevnar 13®, PCV-13

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of the SHAN6™ vaccine to the licensed SHAN5™ given with bOPV and IPV vaccines when coadministered with PCV and ORV

Secondary Objective:

* To describe the immunogenicity profile of the SHAN6™ vaccine 3-dose primary infant vaccination and that of the control vaccines (SHAN5™ given with bOPV and IPV)
* To describe the immune response to co-administered ORV-1 (Rotarix™) in a subset of participants from each group
* To describe the immune response to co-administered PCV-13 (Prevnar 13®) in a subset of participants from each group
* To describe the persistence of the antibodies against SHAN6™ antigens following a 3-dose primary series of SHAN6™ or SHAN5™ given with bOPV and IPV
* To describe the immunogenicity profile of SHAN6™ 28 days after the single booster dose of SHAN6™
* To describe the safety profile of the SHAN6™ vaccine and the control vaccines (SHAN5™ given with bOPV and IPV), when administered concomitantly with routine pediatric vaccines

DETAILED DESCRIPTION:
The duration of each participant's active participation in the study will be approximately 14-17 months (416-506 days)

in addition to the 2 MedDRA terms: Polio immunisation 10054175 Hepatitis B immunisation 10054181 Haemophilus influenzae type B immunisation 10069533 Tetanus immunisation 10054131 Rotavirus immunisation 10076886 Pneumococcal immunisation 10069578

ELIGIBILITY:
Inclusion criteria :

* Aged ≥ 2 months (age range of 8 weeks <12 weeks) on the day of the first vaccination
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg or medically stable prematurely born infants (born after a gestational period of 27-36 weeks)
* Infants who have received the birth dose of Bacille Calmette-Guérin vaccine (BCG) at least 4 weeks before the first trial vaccination
* Participant and parent(s)/legally acceptable representative(s) are able to attend all scheduled visits and comply with all study procedures

Exclusion criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine within the period of 4 weeks before to 4 weeks after each trial vaccination, except for oral polio vaccine (OPV) and influenza vaccination. OPV may be received any time during the study while influenza vaccination may be received at a gap of at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B (except the dose of Hep B vaccine given at birth or at least 4 weeks before the first trial vaccination), Haemophilus influenzae type b, poliomyelitis (except OPV), rotavirus, and Streptococcus pneumoniae with either the trial vaccines or another vaccine
* Receipt of immune globulins, blood or blood-derived products since birth
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy since birth; or long-term systemic corticosteroid therapy (prednisone or equivalent at ≥ 0.5 mg/kg/day for more than 2 consecutive weeks since birth)
* Known personal or maternal history of Human Immunodeficiency Virus (HIV), hepatitis B (HBsAg positive), or hepatitis C (hepatitis C virus [HCV] ribonucleic acid [RNA] positive)
* Individuals with blood dyscrasias, leukemia, lymphoma of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, Haemophilus influenzae type b, rotavirus, or pneumococcal infection(s) confirmed either clinically, serologically, or microbiologically
* History of any neurologic disorders, including encephalopathy, seizures (febrile and non-febrile) and progressive neurologic disorders
* History of intussusception
* In an emergency setting, or hospitalized
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia, as reported by the parent/legally acceptable representative, contraindicating intramuscular vaccination in the Investigator's opinion
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion
* Chronic illness that, in the Investigator's opinion, is at a stage where it might interfere with trial conduct or completion
* Any condition which, in the Investigator's opinion, might interfere with the evaluation of the study objectives
* Moderate or severe acute illness/infection (according to the Investigator's judgment) on the day of vaccination or febrile illness (axillary temperature ≥ 38.0 C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Identified as a natural or adopted child of the Investigator, relatives or employee with direct involvement in the proposed study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 8 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 460 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with antibodies (Ab) above predefined threshold against diphtheria (D), tetanus (T), hepatitis B (Hep B), Haemophilus influenzae type b (Hib) and poliovirus (Polio) antigens | 28 days after the third dose (Day 148)
  Ab titers against D, T, Hep B, Hib and Polio antigens will be measured Threshold values will be considered
Adjusted Geometric Mean Concentrations (aGMCs) of Ab against pertussis antigens | 28 days after the third dose (Day 148)
  Ab against pertussis antigens will be measured

SECONDARY OUTCOMES:
Number of participants with Ab titers above predefined thresholds against each antigen diphtheria, tetanus, hepatitis B, Haemophilus influenzae type b and poliovirus antigens | At baseline (Day 0) and 28 days after the third dose (Day 148)
  Ab titers against D, T, Hep B, Hib and polio antigens will be measured Threshold values will be considered
Number of participants with a vaccine response for pertussis antigens | At baseline (Day 0) and 28 days after the third dose (Day 148)
  Pertussis antigens vaccine response Threshold values will be considered
Pertussis antigens vaccine seroconversion | At baseline (Day 0) and 28 days after the third dose (Day 148)
  Ab against pertussis antigens will be measured
Geometric Mean Concentrations Ratios (GMCRs) of Ab against all the antigens, including anti-rotavirus and anti-S. pneumoniae in a subset of participants | At baseline (Day 0) and 28 days after the third dose (Day 148)
  Ab concentrations against all the antigens, including anti-rotavirus and anti-S. pneumoniae for a subset of participants, will be measured The ratio calculated will be: (post dose 3/pre-primary)
GMCs of Ab against each antigen, including anti-rotavirus and anti-pneumococcal serotypes, in a subset of participants | At baseline (Day 0) and 28 days after the third dose (Day 148)
  Ab concentrations against each antigen, including anti rotavirus and anti pneumococcal serotypes for a subset of participants, will be measured
Number of participants with anti-rotavirus Ab titers above predefined thresholds in a subset of participants | At baseline (Day 0) and 28 days after the third dose (Day 148)
  Ab against rotavirus will be measured in a subset of participants Threshold values will be considered
Number of participants with anti-pneumococcal Ab titers above predefined thresholds in a subset of participants | At baseline (Day 0) and 28 days after the third dose (Day 148)
  Anti-pneumococcal Ab will be measured in a subset of participants Threshold values will be considered
Number of participants with Ab titers above predefined threshold against diphtheria, tetanus, hepatitis B, Haemophilus influenzae type b and poliovirus antigens | Before and 28 days after the booster dose (at Day 388-478 and Day 416-506)
  Ab against D, T, Hep B, Hib and polio antigens will be measured Threshold values will be considered
Number of participants with a booster response for pertussis antigens | Before and 28 days after the booster dose (at Day 388-478 and Day 416-506)
  Pertussis antigens booster response Threshold values will be considered
Pertussis antigens vaccine seroconversion | Before and 28 days after the booster dose (at Day 388-478 and Day 416-506)
  Ab against pertussis antigens will be measured
GMCRs of Ab against all the antigens | Before and 28 days after the booster dose (at Day 388-478 and Day 416-506)
  Ab concentrations against all the antigens will be measured The ratio calculated will be: (post booster/pre-booster)
GMCs of Ab against each antigen | Before and 28 days after the booster dose (at Day 388-478 and Day 416-506)
  Ab concentrations against each antigen will be measured
aGMCs of Ab against pertussis antigens | Before and 28 days after the booster dose (at Day 388-478 and Day 416-506)
  Ab against pertussis antigens will be measured, adjusted for baseline value
Number of participants reporting immediate systemic adverse events (AEs) | Within 30 minutes post-vaccination
  Unsolicited (spontaneously reported) systemic AEs
Number of participants reporting solicited injection site and systemic reactions | Up to 7 days post-vaccination
  Solicited injection site reactions:
  - tenderness, erythema and site swelling
  Solicited systemic reactions:
  - fever, vomiting, crying abnormal, drowsiness, appetite lost and irritability
Number of participants reporting unsolicited non-serious AEs | Up to 28 days post-vaccination
  Unsolicited non-serious AEs
Number of participants reporting serious adverse events (SAEs) | Up to Day 416-506
  SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- Thailand (3):
  - Investigational Site Number 7640003, Bangkok
  - Investigational Site Number 7640001, Bangkok
  - Investigational Site Number 7640002, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Sanchez L, Rungmaitree S, Kosalaraksa P, Jantarabenjakul W, Leclercq J, Yaiprayoon Y, Midde VJ, Varghese K, Mangarule S, Noriega F. Immunogenicity and Safety of a Hexavalent DTwP-IPV-HB-PRP~T Vaccine Versus Separate DTwP-HB-PRP~T, bOPV, and IPV Vaccines Administered at 2, 4, 6 Months of Age Concomitantly With Rotavirus and Pneumococcal Conjugate Vaccines in Healthy Infants in Thailand. Pediatr Infect Dis J. 2023 Aug 1;42(8):711-718. doi: 10.1097/INF.0000000000003975. Epub 2023 Apr 27. PMID 37257121
- See also: SH600009 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25345&tenant=MT_SNY_9011